CLINICAL TRIAL: NCT01806597
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Demonstrate the Efficacy at 16 Weeks of Secukinumab 150 and 300 mg s.c. and to Assess Safety, Tolerability and Long-term Efficacy up to 132 Weeks in Subjects With Moderate to Severe Palmoplantar Psoriasis
Brief Title: Study of Safety, Tolerability, and Efficacy of Secukinumab in Subjects With Moderate to Severe Palmoplantar Psoriasis
Acronym: GESTURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457A2312; 2012-005412-25 (EudraCT Number)
Record Dates: First submitted 2013-01-23; First posted 2013-03-07 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Moderate to Severe Palmoplantar Psoriasis
Keywords: Skin condition, itching, psoriasis vulgaris, relapsing remitting psoriasis, immune-med systemic disease, skin lesions, scaly patches, papules, plaques
MeSH Terms: conditions — Skin Diseases; Pruritus; Plaque, Amyloid | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- secukinumab 150mg (Experimental): 201 subjects were randomized in a 1:1:1 ratio to secukinumab either 150 mg or 300 mg, or placebo. Subjects assigned to secukinumab 150 mg were dosed weekly for the first five weeks, then every four weeks up to and including Week 128. To maintain blinding, subjects received additional placebo injections at Weeks 17, 18 and 19. All doses of study treatment were administered by sub-cutaneous injections.
  Interventions: Biological: secukinumab 150 mg
- secukinumab 300 mg (Experimental): 201 subjects were randomized in a 1:1:1 ratio to secukinumab either 150 mg or 300 mg, or placebo. Subjects assigned to secukinumab 300 mg were dosed weekly for the first five weeks and then every four weeks up to and including Week 128. In order to maintain the blinding, subjects received additional placebo injections at Weeks 17, 18 and 19. All doses of study treatment were administered by sub-cutaneous injections.
  Interventions: Biological: secukinumab 300 mg
- Placebo (Placebo Comparator): 201 subjects were randomized in a 1:1:1 ratio to secukinumab either 150 mg or 300 mg, or placebo. Subjects on placebo were dosed weekly for 5 weeks then once every 4 weeks. At Week 16, ppIGA responders continued to receive placebo weekly for 5 weeks starting at Week 16, then every 4 weeks up to and including Week 76 while ppIGA non-responders were randomized in a 1:1 ratio to secukinumab either 150 mg or 300mg weekly for 5 weeks, starting at Week 16, then every 4 weeks up to and including Week 128. At Week 80, subjects on placebo were either terminated their participation, if ppIGA responders, or randomized in a 1:1 ratio to secukinumab either 150 mg or 300 mg once every 4 weeks until Week 128 inclusive. All doses of study treatment were administered by sub-cutaneous injections.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: secukinumab 150 mg — Study treatment were provided in pre-filled syringes of secukinumab 150 mg in 1 mL. Each dosing consiseds of one secukinumab 150 mg s.c. injection plus one placebo secukinumab s.c. injection and took place once weekly during five weeks (at Baseline, Weeks 1, 2, 3 and 4), then once every four weeks starting at Week 8 until Week 128 inclusive. In order to maintain the blinding, patients also received two placebo injections at Weeks 17, 18 and 19. Patients self-administered study treatment under the supervision of site personnel when injections occur during study visits, or at home otherwise.
  Other Names: AIN457 150 mg
  Arms: secukinumab 150mg
Biological: secukinumab 300 mg — Study treatment were provided in pre-filled syringes of secukinumab 150 mg in 1 mL. Each dosing consisted of two secukinumab 150 mg s.c. injections and took ke place once weekly during five weeks (at Baseline, Weeks 1, 2, 3 and 4), then once every four weeks starting at Week 8 until Week 128 inclusive. In order to maintain the blinding, patients also receives two placebo injections at Weeks 17, 18 and 19. Patients self-administered study treatment under the supervision of site personnel when injections occur during study visits, or at home otherwise.
  Other Names: AIN457 300 mg
  Arms: secukinumab 300 mg
Biological: Placebo — Placebo were provided in 1 mL pre-filled syringes. Each dosing consisted of two s.c. injections and took place once weekly during five weeks (at Baseline, Weeks 1, 2, 3 and 4), then at Week 8 and at Week 12. At Week 16, ppIGA responders continued on placebo with dosing at Weeks 16, 17, 18, 19 and 20, then once every four weeks from Week 24 until Week 76 inclusive. At Week 80, ppIGA responders ended their participation in the study while ppIGA non-responders were re-randomized, to receive 150 mg or 300 mg secukinumab once every four weeks starting at Week 80 until Week 128 inclusive. Patients self-administered study treatment under the supervision of site personnel when injections occur during study visits, or at home otherwise.
  Arms: Placebo

SUMMARY:
Purpose of the study was to demonstrate the efficacy of secukinumab versus placebo on palmoplantar psoriasis and to assess the long term efficacy, safety and tolerability of secukinumab.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic, moderate to severe plaque type psoriasis for at least 6 months prior to randomization and significant involvement of the palms and soles at baseline, defined as palmoplantar Investigator's Global Assessment (ppIGA) score of ≥ 3 on a 5-point scale, as well as at least one skin plaque at baseline which is not in the palmoplantar area
* Candidates for systemic therapy, i.e. psoriasis inadequately controlled by topical treatment (including super potent topical corticosteroids) and/or phototherapy and/or previous systemic therapy

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque type psoriasis (e.g., pustular psoriasis, palmoplantar pustulosis, acrodermatitis of Hallopeau, erythrodermic and guttate psoriasis)
* Drug-induced psoriasis (e.g. new onset or current exacerbation from β-blockers, calcium channel inhibitors or lithium)
* Ongoing use of prohibited treatments (e.g. topical or systemic corticosteroids (CS), UV therapy). Washout periods do apply.
* Prior exposure to secukinumab (AIN457) or any other biological drug directly targeting IL-17 or the IL-17 receptor
* Use of any investigational drugs within 4 weeks prior to study treatment initiation or within a period of 5 half-lives of the investigational treatment, whichever is longer
* Active ongoing inflammatory diseases other than psoriasis that might confound the evaluation of the benefit of secukinumab therapy
* History of hypersensitivity to constituents of the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2013-06-19 (Actual); Primary Completion 2016-11-02 (Actual); Study Completion 2016-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (50):
- United States (8):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Verona, New Jersey
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Goodlettsville, Tennessee
- Australia (4):
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Carlton, Victoria
  - Novartis Investigative Site, East Melbourne, Victoria
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Liège
- Canada (5):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Barrie, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Finland (2):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Tampere
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Szeged
- Israel (3):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Tel Aviv
- Netherlands (3):
  - Novartis Investigative Site, Breda, CK
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Stavanger, Norway
- Portugal (3):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Russia (3):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Slovakia (3):
  - Novartis Investigative Site, Kosice-Saca, Slovak Republic
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Svidník
- Spain (3):
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Las Palmas de Gran Canaria, Las Palmas de G.C
  - Novartis Investigative Site, Barcelona
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Fatih / Istanbul, Turkey
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Gaziantep
- United Kingdom (2):
  - Novartis Investigative Site, London, England
  - Novartis Investigative Site, Dudley, West Midlands

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Week 16 was considered the first dose of Treatment Period 2. Week 132 visit was the final visit of Treatment Period 2, and no study treatment was administered at this visit.
Pre-assignment Details: Patients who completed Period 2 & patients who prematurely discontinued treatment or withdrew from study entered the treatment-free Follow-up (FU) Period (no study treatment was administered during Period) included only 1 visit at Week 140 (End of FU), which was 8 weeks after the end of Period 2 & 12 weeks after the last dose of study drug.
Groups:
- AIN457 150mg: AIN457 150mg sub-cutaneous (s.c.) injection plus a placebo AIN457 s.c. injection once weekly for 5 weeks followed by dosing every 4 weeks
- AIN457 300 mg: AIN457 300 mg (2 s.c. injections of the 150 mg dose) once weekly for 5 weeks followed by dosing every 4 weeks
- Placebo - AIN457 150 mg: all placebo patients who were re-randomized to secukinumab 150 mg at re-randomization
- Placebo - AIN457 300mg: all placebo patients who were re-randomized to AIN457 300 mg at re-randomization
- Placebo: placebo AIN457 (2 sc injections) once weekly for 5 weeks, followed by dosing every 4 weeks.
- Any AIN457 Dose: All patients who were injected with AIN457
Period: Period 1 (Baseline to Week 16)
Arm/Group | AIN457 150mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300mg | Placebo | Any AIN457 Dose
Started | 68 | 69 | 0 | 0 | 68 | 0
Completed | 63 | 64 | 0 | 0 | 63 | 0
Not Completed | 5 | 5 | 0 | 0 | 5 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 2 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 0 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (Week 16 to Week 132)
Arm/Group | AIN457 150mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300mg | Placebo | Any AIN457 Dose
Started | 63 | 64 | 31 | 31 | 1 | 0
Completed | 24 | 44 | 17 | 20 | 0 | 0
Not Completed | 39 | 20 | 14 | 11 | 1 | 0
Not completed — Adverse Event | 9 | 6 | 4 | 3 | 1 | 0
Not completed — Lack of Efficacy | 12 | 5 | 3 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 0 | 0
Not completed — study terminated by sponsor | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 5 | 6 | 5 | 0 | 0
Not completed — non-compliance with study treatment | 2 | 2 | 1 | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0
Period: Follow-up Period (Week 132 to Week 140)
Arm/Group | AIN457 150mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300mg | Placebo | Any AIN457 Dose
Started | 0 | 0 | 0 | 0 | 3 | 161
Completed | 0 | 0 | 0 | 0 | 3 | 149
Not Completed | 0 | 0 | 0 | 0 | 0 | 12
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 150mg | AIN457 300 mg | Placebo | Total
Number analyzed (Participants) | 68 | 69 | 68 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (12.56) | 48.8 (14.21) | 50.9 (12.95) | 50.7 (13.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 31 | 34 | 93
  Male | 40 | 38 | 34 | 112

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Participants With Palmoplantar Investigator Global Assessmnet (ppIGA) 0 or 1 Response After 16 Weeks of Treatment
Description: palmoplantar Investigator's Global Assessment (ppIGA) response after 16 weeks of treatment. To be considered a ppIGA responder at Week 16, a subject must have ppIGA of 0 or 1 at Week 16 and a reduction of at least 2 points on the ppIGA scale from baseline.
Time Frame: Week 16
Population: Full Analysis Set (FAS): The FAS comprised of all patients from the randomized set to who study treatment had been assigned. Following the intent-to-treat principle, patients were analyzed according to the treatment assigned to at randomization.
Measure: Number; unit: Percentages of participants
Arm/Group | AIN457 150mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 68 | 69 | 68
Percentages of participants | 22 | 33.3 | 1.5
Statistical Analysis 1: Comparison: AIN457 150mg vs Placebo; Data at Week 16 was analyzed using the stratified Cochran-Mantel-Haenszel-test. The test was stratified by body-weight category (<90 kg or ≥90 kg); Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 19.3, 95% CI 2-sided [2.4 to 154.6]
Statistical Analysis 2: Comparison: AIN457 300 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 29.4, 95% CI 2-sided [4.1 to 211.9]

2. Secondary Outcome: Percentages of Participants With Palmoplantar Investigator Global Assessment (ppIGA) 0 or 1 Response - Treatment Period I
Description: ppIGA: Palmoplantar Ivestigator's Global Assessment. The IGA mod 2011 rating scale: The IGA mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe.
  Based on this scale, a patient was considered as an IGA 0 or 1 responder if they achieved a score of 0 or 1 and improved by at least 2 points on the IGA scale at a given time point compared to their score at randomization (baseline).
Time Frame: Week 1, week 2, week 4, week, 8, week 12, week 16
Population: FAS
Measure: Number; unit: Percentages of participants
Arm/Group | AIN457 150mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 68 | 69 | 68
Percentages of participants
  Week 1 | 1.5 | 1.4 | 0
  Week 2 | 1.5 | 7.2 | 0
  Week 4 | 4.4 | 8.7 | 0
  Week 8 | 17.6 | 26.1 | 0
  Week 12 | 20.6 | 33.3 | 1.5
  Week 16 | 22.1 | 33.3 | 1.5

3. Secondary Outcome: Percentages of Subjects With ppIGA 0 or 1 Response (Observed Cases) - Treatment Period II
Description: as for outcome 2
Time Frame: Week 16, Week 20, Week 28, Week 32, Week 64, Week 132
Population: FAS
Measure: Number; unit: Percentages of participants
Groups:
- Placebo - AIN457 300 mg: all placebo patients who were re-randomized to secukinumab 300 mg at re-randomization.
- Placebo: Placebo AIN457 (2sc injections) once weekly for 5 weeks followed by dosing every 4 weeks
Arm/Group | AIN457 150mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg | Placebo
Number analyzed (Participants) | 68 | 69 | 31 | 31 | 1
Percentages of participants
  Week 16 | 22.1 (15.624) | 33.3 (12.074) | 0.0 (8.880) | 0.0 (7.983) | 100.0 (4.479)
  Week 20 | 32.4 (14.307) | 33.3 (13.104) | 12.9 (11.570) | 9.7 (12.625) | 0.0 (NA)
  Week 28 | 29.4 (15.232) | 44.9 (14.258) | 32.3 (14.560) | 51.6 (10.441) | 100.0 (NA)
  Week 32 | 29.4 (14.658) | 42.0 (11.688) | 35.5 (11.728) | 41.9 (5.844) | 0.0 (NA)
  Week 64 | 26.5 | 46.4 | 29.0 | 48.4 | 0.0
  Week 132 | 22.1 | 27.5 | 12.9 | 35.5 | 0.0

4. Secondary Outcome: Percentages of Subjects With ppIGA 0 or 1 Response (Observed Cases) - Entire Treatment Period
Description: as for outcome 2
Time Frame: Week 16, Week 24, Week 28, Week 80
Population: FAS
Measure: Number; unit: Percentages of participants
Arm/Group | AIN457 150mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg | Placebo
Number analyzed (Participants) | 68 | 69 | 31 | 31 | 6
Percentages of participants
  Week 16: number analyzed (Participants) | 68 | 69 | 31 | 31 | 4
  Week 16 | 23.4 | 37.7 | 0.0 | 0.0 | 25.0
  Week 24: number analyzed (Participants) | 68 | 69 | 31 | 31 | 1
  Week 24 | 40.7 | 44.1 | 20.0 | 36.7 | 100.0
  Week 28: number analyzed (Participants) | 68 | 69 | 31 | 31 | 1
  Week 28 | 34.5 | 50.8 | 20.0 | 48.3 | 0.0
  Week 80: number analyzed (Participants) | 68 | 69 | 31 | 31 | 0
  Week 80 | 41.7 | 65.3 | 45.0 | 68.2 |

5. Secondary Outcome: Absolute Change From Baseline for Palmoplantar Psoriasis Area and Severity Index (ppPASI) Score -Treatment Period I
Description: Psoriasis Area and Severity Index (PASI) is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease).
Time Frame: Week 1, Week 2, Week 4, Week 8, Week 12, Week 16
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457 150mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 68 | 69 | 68
Units on a scale
  Week 1 | -1.13 (4.797) | -2.22 (4.334) | -0.85 (3.355)
  Week 2 | -3.11 (7.669) | -5.32 (6.120) | -1.90 (5.434)
  Week 4 | -6.69 (9.890) | -9.18 (9.734) | -3.95 (7.424)
  Week 8 | -9.74 (12.779) | -11.30 (11.954) | -3.22 (8.316)
  Week 12 | -10.15 (14.409) | -12.83 (12.286) | -3.07 (8.479)
  Week 16 | -9.41 (15.984) | -13.35 (12.941) | -2.43 (8.527)

6. Secondary Outcome: Absolute Change From Baseline for Palmoplantar Psoriasis Area and Severity Index (ppPASI) Score (Observed Cases) - Entire Treatment Set
Description: as for outcome 5
Time Frame: Week 16, Week 32, Week 80, Week 132
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457 150mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg | Placebo
Number analyzed (Participants) | 68 | 69 | 31 | 31 | 6
Units on a scale
  Week 16: number analyzed (Participants) | 64 | 61 | 30 | 30 | 4
  Week 16 | -8.97 (15.624) | -12.67 (12.074) | -1.57 (8.880) | -3.11 (7.983) | -7.15 (4.479)
  Week 32: number analyzed (Participants) | 52 | 60 | 25 | 29 | 1
  Week 32 | -16.29 (14.307) | -17.43 (13.104) | -15.49 (11.570) | -15.09 (12.625) | -11.40
  Week 80: number analyzed (Participants) | 36 | 49 | 20 | 22 | 0
  Week 80 | -18.05 (15.232) | -19.27 (14.258) | -13.71 (14.560) | -16.70 (10.441) |
  Week 132: number analyzed (Participants) | 21 | 28 | 12 | 18 | 0
  Week 132 | -16.74 (14.658) | -19.16 (11.688) | -17.07 (11.728) | -13.82 (5.844) |

7. Secondary Outcome: Number of Participants Developing Anti-secukinumab Antibodies
Description: To investigate the development of immunogenicity against secukinumab
Time Frame: Over time up to week 132
Population: FAS
Measure: Count of Participants; unit: Participants
Groups:
- Placebo - AIN 150mg: all placebo patients who were re-randomized to AIN457 150 mg at re-randomization
Arm/Group | AIN457 150mg | AIN457 300 mg | Placebo - AIN 150mg | Placebo - AIN457 300mg
Number analyzed (Participants) | 68 | 69 | 31 | 31
Participants | 2 | 2 | 2 | 3

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First treatment until Last Patient Last Visit.
Groups:
- Any AIN457 150 mg: AIN457 150mg subcutaneous (s.c.) injection plus a placebo AIN457 s.c. injection once weekly for 5 weeks followed by dosing every 4 weeks
- Any AIN457 300 mg: AIN457 300mg subcutaneous ((2 s.c. injections of the 150 mg dose) once weekly for 5 weeks followed by dosing every 4 weeks
Arm/Group | Any AIN457 150 mg | Any AIN457 300 mg | Placebo | Any AIN457 Dose
Serious Adverse Events (participants affected / at risk) | 19/99 | 13/100 | 2/68 | 32/199
Other Adverse Events (participants affected / at risk) | 75/99 | 68/100 | 30/68 | 143/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg (N=99) | Any AIN457 300 mg (N=100) | Placebo (N=68) | Any AIN457 Dose (N=199)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1
Infective keratitis (Infections and infestations) | 1 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Peripheral nerve injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0 | 1
Transient global amnesia (Nervous system disorders) | 1 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 3
Miscarriage of partner (Social circumstances) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg (N=99) | Any AIN457 300 mg (N=100) | Placebo (N=68) | Any AIN457 Dose (N=199)
Blepharitis (Eye disorders) | 2 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 1 | 4
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 3
Dental caries (Gastrointestinal disorders) | 2 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 0 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 3 | 1 | 6
Nausea (Gastrointestinal disorders) | 3 | 1 | 0 | 4
Toothache (Gastrointestinal disorders) | 2 | 2 | 0 | 4
Chills (General disorders) | 2 | 0 | 0 | 2
Fatigue (General disorders) | 4 | 1 | 0 | 5
Influenza like illness (General disorders) | 1 | 3 | 0 | 4
Injection site haematoma (General disorders) | 2 | 1 | 0 | 3
Injection site reaction (General disorders) | 2 | 0 | 0 | 2
Oedema peripheral (General disorders) | 5 | 4 | 0 | 9
Peripheral swelling (General disorders) | 2 | 0 | 1 | 2
Pyrexia (General disorders) | 4 | 1 | 0 | 5
Hepatic steatosis (Hepatobiliary disorders) | 2 | 1 | 0 | 3
Bronchitis (Infections and infestations) | 2 | 2 | 1 | 4
Cellulitis (Infections and infestations) | 2 | 2 | 0 | 4
Conjunctivitis (Infections and infestations) | 2 | 3 | 0 | 5
Folliculitis (Infections and infestations) | 2 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 5 | 4 | 0 | 9
Genital infection fungal (Infections and infestations) | 2 | 0 | 0 | 2
Impetigo (Infections and infestations) | 2 | 0 | 0 | 2
Influenza (Infections and infestations) | 4 | 7 | 4 | 11
Localised infection (Infections and infestations) | 0 | 3 | 0 | 3
Nasopharyngitis (Infections and infestations) | 14 | 8 | 4 | 22
Oral candidiasis (Infections and infestations) | 0 | 5 | 0 | 5
Oral herpes (Infections and infestations) | 3 | 2 | 1 | 5
Pharyngitis (Infections and infestations) | 3 | 6 | 0 | 9
Rhinitis (Infections and infestations) | 2 | 2 | 0 | 4
Sinusitis (Infections and infestations) | 1 | 3 | 0 | 4
Skin infection (Infections and infestations) | 2 | 2 | 1 | 4
Tinea pedis (Infections and infestations) | 5 | 1 | 0 | 6
Tonsillitis (Infections and infestations) | 1 | 3 | 0 | 4
Tooth abscess (Infections and infestations) | 2 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 10 | 20 | 3 | 30
Urinary tract infection (Infections and infestations) | 3 | 7 | 0 | 10
Viral upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Muscle strain (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 4
Procedural pain (Injury, poisoning and procedural complications) | 1 | 4 | 0 | 5
Weight increased (Investigations) | 2 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 4 | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 10 | 2 | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 2 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1 | 6
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 4
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 2
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 3
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 0 | 4
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 1
Headache (Nervous system disorders) | 10 | 11 | 6 | 21
Paraesthesia (Nervous system disorders) | 2 | 1 | 0 | 3
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 2
Depression (Psychiatric disorders) | 2 | 1 | 0 | 3
Nephrolithiasis (Renal and urinary disorders) | 3 | 2 | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 4
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 3
Eczema (Skin and subcutaneous tissue disorders) | 4 | 2 | 1 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 4
Psoriasis (Skin and subcutaneous tissue disorders) | 12 | 11 | 4 | 23
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 4
Skin mass (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 4
Haematoma (Vascular disorders) | 2 | 0 | 0 | 2
Hypertension (Vascular disorders) | 5 | 3 | 0 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.